CLINICAL TRIAL: NCT01168050
Title: Phase II Multicentric Uncontrolled National Trial Assessing the Efficacy of Nilotinib in First or Second Line Treatment of Primary Melanomas , Stage III Unresectable Melanomas, or Stage IV Melanomas With c-KIT Mutation or Amplification.
Brief Title: Efficacy of Nilotinib in First or Second Line Treatment of Primary Melanomas Stage III Unresectable Melanomas.
Acronym: NILOMEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia Idir, Department Clinical Research of Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P081237
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Malignant Skin Melanoma T0; Stage III Melanoma; Stage IV Melanoma; Amplification
Keywords: Malignant Skin Melanoma T0; stage III unresectable melanomas,; or stage IV melanomas with c-KIT mutation; or amplification.
MeSH Terms: conditions — Melanoma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 400 mg twice per day

SUMMARY:
NILOMEL is a phase II multicentric uncontrolled open national trial assessing the efficacy of Nilotinib in first or second line treatment of primary melanomas , stage III unresectable melanomas, or Stage IV melanomas with c-KIT mutation or amplification. The primary objective is overall response rate (partial and complete response) according to RECIST 1.1 criteria, assessed using CT-SCAN (stage IV melanoma) or MRI (unresectable melanoma) after 6 months therapy with Nilotinib 800 mg/d. Secondary objectives include:

* Disease control rate (complete, partial response and stable disease)
* Metabolic response
* Tolerance NCI CTCAE Version 3.0
* Biomarkers associated to response and disease control.

DETAILED DESCRIPTION:
NILOMEL is a phase II multicentric uncontrolled open national trial assessing the efficacy of Nilotinib in first or second line treatment of primary melanomas , stage III unresectable melanomas, or Stage IV melanomas with c-KIT mutation or amplification (in case of c-KIT amplification, no B-RAF nor N-Ras mutation should be detected). The primary objective is overall response rate (partial and complete response) according to RECIST 1.1 criteria, assessed using CT-SCAN (stage IV melanoma) or MRI (unresectable melanoma) after 6 months therapy with Nilotinib 800 mg/d. Secondary objectives include:

* Disease control rate (complete, partial response and stable disease) according to RECIST
* Metabolic response rate (TEP-SCAN)
* Tolerance NCI CTCAE Version 3.0
* Biomarkers associated to response and disease control (evaluated at M0, M1 and M6). Protein analysis of c-KIT, PI3K, MAPK and STAT signalling pathways as well as PDGFR and Ephrin signalling pathways.

Patients with progressive disease after 3 months therapy will be withdrawn. Patient with stable disease after 3 months will continue Nilotinib until evaluation at 6 months. Patients with stable disease or progressive disease at 6 months will continue Nilotinib until progression.

The trial has been planned using a one-stage design (Fleming TR) . We considered that a response rate under 7.5% would define the null hypothesis of no efficacy . To detect a response rate of 30% or more with power 90% using a one-sided test at the 0.05 level, 25 patients have to be recruited.

Accrual for 2.5 years total study duration: 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven melanoma with either c-KIT mutation or C-KIT amplification (without BRAF or NRAS mutation)
* Unresectable primary or stage III or stage IV melanoma
* Measurable disease (RECIST)
* The inclusion of patients with primary tumor or metastasis accessible to sequential biopsies will be favored. If such lesions are present, biopsies are mandatory and not optional
* No more than 1 previous specific therapy excluding tyrosine kinase inhibitors. 4 weeks wash out will be needed after cytotoxic therapy , 12 weeks wash out after anti -CTLA4 therapy or any immunological treatment
* No radiotherapy within 4 weeks ; previously irradiated lesion will not be considered as measurable unless progression at inclusion
* ECOG performance status < 2
* WBC ≥ 3,000/mm³
* PNN ≥ 1,500/mm³ (G-CSF allowed)
* platelets ≥ 100,000/mm³
* Hb ≥ 9.0 g/dL ( transfusions allowed as well as recombinant erythropoetin)
* Creatinin clearance > 40ml/mn
* Normal kalemia
* Normal magnesemia
* Total bilirubin <1.5N ; ASAT and ALAT <2.5N
* PT/INR and PTT normal
* NYHA class < 3
* Signed Written Informed Consent
* Affiliated to the National Health Insurance

Exclusion Criteria:

* Patients refusal
* Age < 18 years
* Fertile women who do not want or cannot use effective contraception during the study and up to 8 weeks after the end of study
* Women pregnant or nursing
* Women with positive pregnancy test at inclusion or before treatment initiation
* Fertile and sexually active men whose partner are fertile women who do not use effective contraception
* Clinical and/or radiographic evidence of active cerebral metastases
* Severe evolutive infection
* Known HIV infection
* Concomitant therapy with any other anti-cancer, immunomodulator or immunosuppressing agent or radiotherapy (except palliative care if bone metastases, after acceptance of principal investigator).
* Previous use of tyrosine kinase inhibitors
* More than one line of prior systemic therapies of melanoma by anti-cancer agent or immunotherapy.
* Received experimental treatment within 4 weeks of inclusion
* Pace-maker
* Cardiac dysfunction, as evaluated by one of:

  * Ejection fraction < 45% (less than 28 days from inclusion)
  * Congenital prolonged QT
  * QTc > 450 ms
  * Ventricular tachyarrhythmia within the past 6 months
  * Bradycardia at rest < 50/mn
  * Major conduction dysfunction
  * Myocardial infarction within the previous 6 months
  * Unstable angina
* Uncontrolled hypertension
* Digestive disease that may inhibited NILITINIB absorption
* Concomitant medication that may increase QT
* Taking CYP3A4 inhibitors
* Eating Sevilla oranges (or Sevilla oranges derivates), grapefruit (or grapefruit juice), grapes (or grapes juice), pomegranate (or pomegranate juice)
* Hereditary galactose intolerance, Lapp-lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Objective response | 6 months
  Partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Disease control | 6 months
  Complete or partial response or stable disease per Response Evaluation Criteria in Solid Tumors (RECIST).
Objective response | 3 months
  Partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST).
Metabolic response | 6 months
  Metabolic response as evaluated by TEP-SCAN
Tolerance | 1 year
  Tolerance will be evaluated according to National Cancer Institute (NCI) Criteria for Adverse Events, CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Lebbe, MD, PhD, Principal Investigator — Hôpital Saint-Louis, Paris, France
Locations (1):
- Hôpital Saint-Louis, Paris, France